CLINICAL TRIAL: NCT02619201
Title: Comparison of Efficacy of Ondansetron Versus Metoclopramide for Vomiting in Children With Acute Gastroenteritis: Randomized Controlled Clinical Trial
Brief Title: Antiemetic Efficacy of Ondansetron Versus Metoclopramide
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital General Naval de Alta Especialidad - Escuela Medico Naval (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HGNAE-10
Record Dates: First submitted 2015-11-25; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-10

CONDITIONS: Acute Gastroenteritis; Vomiting
Keywords: vomiting in children; ondansetron; metoclopramide; antiemetics
MeSH Terms: conditions — Vomiting | interventions — Ondansetron; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ondansetron (Experimental): An intravenous dose of ondansetron ( 0.15mg /kg / doses ) Diluted in 20 ml of saline and administer intravenously in 5 minutes
  Interventions: Drug: Ondansetron
- metoclopramide (Active Comparator): An intravenous dose of metoclopramide ( 0.15mg /kg / doses ) Diluted in 20 ml of saline and administer intravenously in 5 minutes
  Interventions: Drug: metoclopramide

INTERVENTIONS:
Drug: Ondansetron — An intravenous dose of ondansetron ( 0.15mg /kg / doses ) .
  Other Names: OD
  Arms: ondansetron
Drug: metoclopramide — An intravenous dose of metoclopramide ( 0.15mg /kg / doses ) .
  Other Names: MT
  Arms: metoclopramide

SUMMARY:
Acute gastroenteritis (GEA) is a public health problem at present, the main cause of vomiting and consultation in emergencies in children under 5 years. Worldwide, there are about 2 million deaths per year due to gastroenteritis in children under 5 years.

In Mexico, the mortality rate by age in 2013, recorded 28 deaths per 100,000 boys and girls, in 2013 in our country 2.5 million children between 5 and 17 years engaged in an economic activity. The occupancy rate for the child population was 8.6: 11.4 for boys and 5.8 for girls.

NICE guidance gastroenteritis defined as a transient disorder caused by an enteric infection and characterized by a sudden onset of diarrhea with or without vomiting

DETAILED DESCRIPTION:
It will be conducted a randomized controlled double-blinded study in the Emergency service of the Naval General Hospital of High Specialty in the Mexico City. The period of patient inclusion in the study is November 2015 to November 2016.

The selections of the patients are children between 1 and 5 years who come to the emergency room with symptoms of acute gastroenteritis with vomiting and intolerance of oral route.

Treatments were randomly assigned eligible patients on admission in the emergency department

The primary endpoint was evaluated at 15 minutes after treatment application:

* Treatment 1: Ondansetron was administered intravenous dose (0.15mg/kg/doses) Diluted in 20 ml saline and administered intravenously 5 minutes
* Treatment 2: Metoclopramide was administered intravenous dose (0.15mg/kg/doses) Diluted in 20 ml saline and administered intravenously 5 minutes

The administration of intravenous medications, will be held in the observation area of the emergency department of pediatrics under monitoring continuo vital signs during application and 15 minutes after treatment.

At 15 minutes after administration, the mouth with oral electrolyte begins by assessing your tolerance, 30 minutes to progress to the astringent diet.

It will follow up with patient assessment in the emergency department of pediatrics, 3 hours after having established the treatment, in order to corroborate the remission of vomiting, it is graduation of home otherwise he will enter hospital.

Primary objective Cumulative rate of cessation of vomiting

secondary objectives

* Compare the number of vomiting episodes with the administration of ondansetron vs metoclopramide
* Compare time duration in which the oral route is restarted.
* Compare hospital admission rate
* Describe adverse effects in both groups

Inclusion Criteria:

* Orally intolerance
* More than 2 vomiting in the last 24 hours
* Without antiemetic therapy within 24 hours of the clinical picture
* Patients with or without diarrhea

Exclusion Criteria:

* Previous abdominal surgery
* Suspected surgical abdominal
* vomiting bile
* Hypersensitivity to Ondansetron and Metoclopramide

ELIGIBILITY:
Inclusion Criteria:

* Orally intolerance
* More than 2 vomiting in the last 24 hours
* Without antiemetic therapy within 24 hours of the clinical picture
* Patients with or without diarrhea

Exclusion Criteria:

* Previous abdominal surgery
* Suspected surgical abdominal
* Vomiting bile
* Hypersensitivity to Ondansetron and Metoclopramide

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-05 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Cumulative rate of vomiting after cessation of drug administration | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yaneth Miranda Tecuautzin, medicine, Principal Investigator — Secretaria de Marina-Armada de México (Mexican Navy)

REFERENCES:
- [Background] Herikstad H, Yang S, Van Gilder TJ, Vugia D, Hadler J, Blake P, Deneen V, Shiferaw B, Angulo FJ. A population-based estimate of the burden of diarrhoeal illness in the United States: FoodNet, 1996-7. Epidemiol Infect. 2002 Aug;129(1):9-17. doi: 10.1017/s0950268801006628. PMID 12211601
- [Background] Guarino A, Albano F, Ashkenazi S, Gendrel D, Hoekstra JH, Shamir R, Szajewska H; ESPGHAN/ESPID Evidence-Based Guidelines for the Management of Acute Gastroenteritis in Children in Europe Expert Working Group. European Society for Paediatric Gastroenterology, Hepatology, and Nutrition/European Society for Paediatric Infectious Diseases evidence-based guidelines for the management of acute gastroenteritis in children in Europe: executive summary. J Pediatr Gastroenterol Nutr. 2008 May;46(5):619-21. doi: 10.1097/MPG.0b013e31816e219e. No abstract available. PMID 18493225
- [Background] Haque KN, al-Frayh A, el-Rifai R. Is it necessary to regraduate milk after acute gastroenteritis in children? Trop Geogr Med. 1983 Dec;35(4):369-73. PMID 6689452
- [Background] Carter B, Fedorowicz Z. Antiemetic treatment for acute gastroenteritis in children: an updated Cochrane systematic review with meta-analysis and mixed treatment comparison in a Bayesian framework. BMJ Open. 2012 Jul 19;2(4):e000622. doi: 10.1136/bmjopen-2011-000622. Print 2012. PMID 22815462
- [Background] National Collaborating Centre for Women's and Children's Health (UK). Diarrhoea and Vomiting Caused by Gastroenteritis: Diagnosis, Assessment and Management in Children Younger than 5 Years. London: RCOG Press; 2009 Apr. Available from http://www.ncbi.nlm.nih.gov/books/NBK63844/ PMID 22132432
- [Background] Atia AN, Buchman AL. Oral rehydration solutions in non-cholera diarrhea: a review. Am J Gastroenterol. 2009 Oct;104(10):2596-604; quiz 2605. doi: 10.1038/ajg.2009.329. Epub 2009 Jun 23. PMID 19550407
- [Background] Freedman SB, Adler M, Seshadri R, Powell EC. Oral ondansetron for gastroenteritis in a pediatric emergency department. N Engl J Med. 2006 Apr 20;354(16):1698-705. doi: 10.1056/NEJMoa055119. PMID 16625009
- [Background] Rerksuppaphol S, Rerksuppaphol L. Randomized study of ondansetron versus domperidone in the treatment of children with acute gastroenteritis. J Clin Med Res. 2013 Dec;5(6):460-6. doi: 10.4021/jocmr1500w. Epub 2013 Oct 12. PMID 24171058
- [Background] Das JK, Kumar R, Salam RA, Freedman S, Bhutta ZA. The effect of antiemetics in childhood gastroenteritis. BMC Public Health. 2013;13 Suppl 3(Suppl 3):S9. doi: 10.1186/1471-2458-13-S3-S9. Epub 2013 Sep 17. PMID 24564795
- [Background] Roslund G, Hepps TS, McQuillen KK. The role of oral ondansetron in children with vomiting as a result of acute gastritis/gastroenteritis who have failed oral rehydration therapy: a randomized controlled trial. Ann Emerg Med. 2008 Jul;52(1):22-29.e6. doi: 10.1016/j.annemergmed.2007.09.010. Epub 2007 Nov 19. PMID 18006189